CLINICAL TRIAL: NCT03764176
Title: Accuracy of Computer-assisted Template-based Implant Placement Using Conventional Impression and Scan Model or Digital Impression: a Randomized Controlled Trial
Brief Title: Accuracy of Computer-assisted Template-based Implant Placement Using Conventional or Digital Impression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Peñarrocha Oltra, Assistant Postdoctoral Lecturer (Profesor Ayudante Doctor), University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H1497613138277
Record Dates: First submitted 2018-11-27; First posted 2018-12-04 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Dental Implant Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional impression (Active Comparator): The intervention of this arm will be "conventional impression": polyether impression will be taken with a customized tray.
  Interventions: Procedure: Conventional impressions
- Digital impression (Experimental): The intervention of this arm will be "digital impression": digital impression will be taken using a CS 3600 intraoral scanner .
  Interventions: Procedure: Digital impressions

INTERVENTIONS:
Procedure: Conventional impressions — In the conventional group, a polyether impression (ImpregumTM, 3M ESPE, Seefeld, Germany) will be taken with a customized tray (Diatray Top, Dental Kontor, Stockelsdorf, Germany). The impression will be poured with Gypsum IV Class Scale 5° (T6, Techim, Techim Group s.r.l., Arese, Italy) and then, the models mounted in a fully adjustable articulator (Protar Evo 7, KaVo Dental, Biberach, Germany). Afterwards, a dental wax-up will be made accordingly to the functional and esthetic requirements. Finally, master model and wax-up will be digitalized by using a lab scanner.
  A surgical template will be derived from the mounted casts (conventional group) and used to place the implants using guided surgery.
  Arms: Conventional impression
Procedure: Digital impressions — Patients will be randomly assigned to undergo intraoral digital impression (digital group) or conventional impression (conventional group). In the digital group, a digital impression will be taken using CS 3600 intraoral scanner (Carestream Dental LLC, Atlanta, GA, USA). The digital data (STL, STereo Lithography interface format) will be imported in a 3D design software to realize a virtual wax-up according to the functional and esthetic requirements.
  A surgical template will be derived from the virtual plane (digital group) and used to place the implants using guided surgery.
  Arms: Digital impression

SUMMARY:
Proper implant position has a significant impact in esthetic and functional outcomes of implant-supported restorations. Computer-assisted template-based implant placement (guided surgery) have become increasingly popular due to improved planning and the higher transfer accuracy of the virtual plan to the surgical site compared with freehand insertion or freehand final drilling. Digital impressions replace the need for traditional materials that can be inconvenient and messy for patients. To the best of our knowledge, at the time of planning this study, there were no published RCTs evaluating a fully digital approach for computer-assisted template-based implant placement.

The aim of the present study is to compare early implant failure, template-related complications, and virtual planning accuracy of computer-assisted template-based implant placement using conventional impression and scan model or digital impression.

The null hypothesis is that there will be no difference between these interventions.

ELIGIBILITY:
Inclusion Criteria:

* fully or partially edentulous patient, aged 18 years or older, able to sign an informed consent, in need of an implant-supported fixed restoration will be considered eligible for this study. Any potential implant locations based on individual patient requirements will be considered eligible in the present trial. No set location or group of locations will be excluded.

Exclusion Criteria:

* general medical contraindication to oral surgery (American Society of Anesthesiologist, ASA, class III or IV); irradiation in the head and neck area less than one year before implantation; psychiatric problems; alcohol or drug abuse; pregnant or nursing; untreated periodontitis; severe bruxism or clenching; uncontrolled diabetes; poor oral hygiene and motivation; and inability to complete the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Linear distance between planned and real implant apex position | Immediate post-surgery
  The change in mm between the apex of the planned and the final (real) position of the implant.
Angle between the planned and real implant axis | Immediate post-surgery
  Change in angulation between the planned and the final (real) position of the implant.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Odontológica de la Universitat de Valencia, Fundación Lluis Alcanyis, Valencia, Spain